CLINICAL TRIAL: NCT02152345
Title: A Randomized Clinical Trial of Efficacy and Safety on the Use of Belatacept as Compared to Tacrolimus in the Setting of Rabbit Antithymocyte Globulin Induction and Rapid Steroid Discontinuation in Deceased Donor Renal Transplant Recipients With a Focus on Ameliorating Delayed Graft Function
Brief Title: Belatacept Compared to Tacrolimus in Deceased Donor Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Mark A Hardy, Auchincloss Professor of Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAL7011
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Implant or Graft; Rejection
Keywords: kidney; renal; transplant; belatacept; delayed graft function; thymoglobulin; tacrolimus; kidney function; immunosuppression; NGAL
MeSH Terms: conditions — Rejection, Psychology; Delayed Graft Function | interventions — Abatacept; Tacrolimus; Mycophenolic Acid; Neoadjuvant Therapy; Antilymphocyte Serum; Methylprednisolone; Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Belatacept Immunosuppression (Experimental): Renal transplant recipients will receive steroids (Methylprednisolone), rATG, Belatacept and Mycophenolate. Subjects will be followed for primary endpoint to Day 7 and Month 3 after transplantation and secondary endpoints of kidney function and patient and graft survival up to month 36 after transplantation.
  Interventions: Drug: Belatacept; Drug: Mycophenolate; Drug: rATG; Drug: Methylprednisolone; Procedure: Renal transplant
- Standard Immunosuppression (Tacrolimus) (Active Comparator): Renal transplant recipients will receive standard immunosuppressive therapy, including steroids (Methylprednisolone), rATG, Tacrolimus and Mycophenolate. Subjects will be followed for primary endpoint to Day 7 and Month 3 after transplantation and secondary endpoints of kidney function and patient and graft survival up to month 36 after transplantation.
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate; Drug: rATG; Drug: Methylprednisolone; Procedure: Renal transplant

INTERVENTIONS:
Drug: Belatacept — Belatacept 10 mg/kg will be administered in the operating room approximately 1 hour prior to kidney allograft reperfusion (Day 0). It will then be administered at 10 mg/kg on the following post-transplantation days: Day 5, 14, 30, 56, and 84.
  Belatacept 5 mg/kg will be administered every four weeks thereafter until end of study.
  Other Names: Nulojix
  Arms: Belatacept Immunosuppression
Drug: Tacrolimus — Tacrolimus 0.05 mg/kg by mouth every 12 hours will be on Day 0 after transplantation. It will then be administered at 8-12 ng/mL on the following post-transplantation days: Day 3-90; at 8-10 ng/mL Day 91-180.
  Tacrolimus 6 - 8 ng/mL will be administered daily thereafter until end of study.
  (standard of care)
  Other Names: Prograf
  Arms: Standard Immunosuppression (Tacrolimus)
Drug: Mycophenolate — An immunosuppressive agent used with other medicines to lower the body's natural immunity in patients who receive kidney transplants.
  720 mg by mouth every 12 hours (Day 0)(1080 mg AA).
  (standard of care)
  Other Names: Myfortic
Drug: rATG — 1.5 mg/kg IV daily on Day 0-3.
  (standard of care)
  Other Names: induction with rabbit anti-thymocyte globulin
Drug: Methylprednisolone — 500 mg (Day 0), 250mg (Day 1), 125mg (Day 2), 75 mg (Day 3) IV administered from Day 0-3.
  (standard of care)
  Other Names: Medrol
Procedure: Renal transplant — Standard organ transplant of a kidney into a patient with end-stage renal disease.
  Other Names: Kidney transplant

SUMMARY:
The main purpose of this study is to ﬁnd out whether treatment to prevent kidney rejection with belatacept in presence of Thymoglobulin induction and withdrawal of steroids will result in less delayed graft function or "sleepy kidney" after transplant than that seen in patients who get tacrolimus as their main drug to prevent rejection instead of belatacept. The investigators will also look at whether patients who get belatacept have the same, lesser or more problems that those who get tacrolimus.

DETAILED DESCRIPTION:
New York Presbyterian Hospital-Columbia University Medical Center (NYPH-CUMC) performs nearly 250 renal transplants annually; of these approximately half are recipients of a variety of deceased donor kidneys, usually with cold ischemia time (CIT) >24 hours leading to an approximate incidence of delayed graft function (DGF) of 50%. The main focus of this study will be to determine whether initial immunosuppression with belatacept with Thymoglobulin induction will result in lower incidence and/or more rapid disappearance of DGF than that observed in patients who receive tacrolimus based immunosuppression. NGAL determinations will bne made in the first months after transplantation to correlate with clinical DGF.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have known Epstein-Barr virus (EBV) serostatus, and that status must be positive
* Adult patients ≥18 years of age, receiving a deceased donor kidney transplant at Columbia University Medical Center (CUMC)
* Patients with a PRA ≤ of 50
* Primary or re-transplant candidates (no more than 5th renal transplant)
* Deceased donor renal transplant recipients
* Candidates eligible for rATG induction
* Patients fully consented prior to transplantation
* Women of reproductive age who are willing to delay pregnancy for the duration of the study and use appropriate recommended contraception

Exclusion Criteria:

* Seronegative or unknown EBV serologic status (due to the risk of post-transplant lymphoproliferative disorder, PTLD), predominantly involving the central nervous system.
* Patients with tuberculosis who have not been treated for latent infection.
* Scheduled to undergo multi-organ transplantation
* Recipients of previous non-renal organ transplant
* Patient receiving 5th renal transplant at the time of screening.
* Patients with a PRA > 50
* Recipient is pre-emptive status.
* Recipient with positive flow crossmatch.
* History or known HIV
* Known hypersensitivity or contra-indications to Belatacept, Tacrolimus, Mycophenolate mofetil (cellcept), or mycophenolic acid
* Use of an investigational drug in the past 30 days before day of surgery
* Enrolled in a clinical trial other than the current
* Lactating or pregnant women
* Donor specific antibodies (DSA) identified at the time of transplantation
* ABO incompatible renal transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Hardy, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients called into the hospital for potential renal transplants were approached for possible participation in the study if they agreed to discuss research and were eligible per study criteria. Patients were given the option to participate or decline.
Groups:
- Belatacept Immunosuppression: Renal transplant recipients will receive Methylprednisolone, rATG, Belatacept and Mycophenolate. Subjects will be followed for primary endpoint to Day 7 and Month 3 after transplantation and secondary endpoints of kidney function and patient and graft survival up to month 36 after transplantation.
  Belatacept 10 mg/kg will be administered in the operating room ~1 hr prior to kidney allograft reperfusion (Day 0). It will then be administered at 10 mg/kg on the following post-transplantation days: 5, 14, 30, 56, & 84.
  Belatacept 5 mg/kg will be administered every four weeks thereafter until end of study.
  Standard of Care:
  * Mycophenolate: 720 mg by mouth every 12 hours (Day 0)(1080 mg AA).
  * rATG: 1.5 mg/kg IV daily on Day 0-3.
  * Methylprednisolone: 500 mg (Day 0), 250mg (Day 1), 125mg (Day 2), 75 mg (Day 3) IV administered Day 0-3.
- Standard Immunosuppression (Tacrolimus): Renal transplant recipients will receive standard immunosuppressive therapy, including steroids (Methylprednisolone), rATG, Tacrolimus and Mycophenolate. Subjects will be followed for primary endpoint to Day 7 and Month 3 after transplantation and secondary endpoints of kidney function and patient and graft survival up to month 36 after transplantation.
  Tacrolimus 0.05 mg/kg PO every 12 hrs will be on Day 0 after transplantation. It will then be administered on the following post-transplantation days: 3-90 at 8-12ng/mL; Day 91-180 at 8-10 ng/mL.
  Standard of Care:
  * Tacrolimus 6 - 8 ng/mL administered daily thereafter until end of study.
  * Mycophenolate: 720 mg by mouth every 12 hours (Day 0)(1080 mg AA).
  * rATG: 1.5 mg/kg IV daily on Day 0-3.
  * Methylprednisolone: 500 mg (Day 0), 250mg (Day 1), 125mg (Day 2), 75 mg (Day 3) IV administered from Day 0-3.
Period: Overall Study
Arm/Group | Belatacept Immunosuppression | Standard Immunosuppression (Tacrolimus)
Started | 28 (The first subject randomized to Belatacept was on 15-Sep-2014.) | 29 (The first subject randomized to Standard Immunosuppression was on 14-Jun-2014.)
Completed | 24 (The last subject randomized to Belatacept was on 29-Dec-2016.) | 24 (The last subject randomized to Standard Immunosuppression was on 25-Dec-2016.)
Not Completed | 4 | 5
Not completed — Case Cancellations | 2 | 4
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belatacept Immunosuppression | Standard Immunosuppression (Tacrolimus) | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 25 | 46
  >=65 years | 7 | 4 | 11
Age, Continuous [Mean (Full Range); unit: years] | 57.4 [42 to 77] | 53.8 [23 to 67] | 55.6 [23 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 25 | 39
  Male | 14 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Delayed Graft Function (DGF)
Description: To assess whether treatment with Thymoglobulin induction and belatacept based maintenance immunosuppression would reduce delayed graft function (DGF) rates among recipients of deceased donor renal transplants as measured by clinical findings and NGAL marker, as specified below and defined by others. This will be compared to the incidence of DGF in patients treated with a Tacrolimus based regimen.
  Patients who require hemodialysis in the first 7 days after transplantation and/or patients whose serum creatinine decreases <10% during 3 consecutive days after the transplant will be considered to have DGF in the absence of other confounding factors such as obstruction or infection. NGAL will be used as a verification marker of DGF.
Time Frame: Up to 3 months post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept Immunosuppression | Standard Immunosuppression (Tacrolimus)
Number analyzed (Participants) | 24 | 24
Participants | 12 | 15

2. Secondary Outcome: Percentage of Participants With Allograft Survival
Description: Allograft survival is defined as functioning renal transplant.
Time Frame: Up to 1 year post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept Immunosuppression | Standard Immunosuppression (Tacrolimus)
Number analyzed (Participants) | 24 | 24
Participants | 24 | 21

3. Secondary Outcome: Number of Participants With an Allograft Rejection Episode
Description: All rejection episodes will be confirmed by renal transplant biopsy provoked by change in renal function not explained by other clinical causes.
Time Frame: Up to 1 year post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept Immunosuppression | Standard Immunosuppression (Tacrolimus)
Number analyzed (Participants) | 24 | 24
Participants | 7 | 11

4. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: Estimated glomerular filtration rate (eGFR) is based on a blood sample (serum creatinine value), age, race, and gender. eGFR estimates best the function of the kidney at any one time.
Time Frame: Up to 1 year post-transplantation
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Belatacept Immunosuppression | Standard Immunosuppression (Tacrolimus)
Number analyzed (Participants) | 24 | 24
mL/min/1.73m^2 | 46 (15.85) | 41 (11.45)

ADVERSE EVENTS:
Arm/Group | Belatacept Immunosuppression | Standard Immunosuppression (Tacrolimus)
All-Cause Mortality (participants affected / at risk) | 4/24 | 1/24
Serious Adverse Events (participants affected / at risk) | 14/24 | 15/24
Other Adverse Events (participants affected / at risk) | 5/24 | 3/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept Immunosuppression (N=24) | Standard Immunosuppression (Tacrolimus) (N=24)
Delayed Graft Function (Renal and urinary disorders) | 12 | 15
Rejection (Renal and urinary disorders) | 7 | 11
EBV quant+ (Infections and infestations) | 3 | 3
CMV quant+ (Infections and infestations) | 9 | 5
BK quant+ (Infections and infestations) | 6 | 3
Posttransplant lymphoproliferative disease (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept Immunosuppression (N=24) | Standard Immunosuppression (Tacrolimus) (N=24)
Bleeding (Blood and lymphatic system disorders) | 5 | 3
Anemia (Blood and lymphatic system disorders) | 3 | 2
Urinary Tract Infection (Renal and urinary disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No